CLINICAL TRIAL: NCT04319952
Title: A Study to Demonstrate the Accuracy of the Femoral Neck Resection Compared to the Selected OPS™ Plan Using the Direct Anterior Approach (DAA)
Brief Title: OPS™ With Direct Anterior Approach (DAA)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corin (Industry)
Responsible Party: Sponsor
Other Study IDs: CSP2019-02
Record Dates: First submitted 2020-03-22; First posted 2020-03-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Primary Total Hip Arthroplasty
Keywords: femoral neck resection; offset; leg length; femoral anteversion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Primary Total Hip Replacement with Metafix™ femoral stem and Trinity™ acetabular cup or TriFit-CF™/TriFit-TS™ femoral stem and Trinity™ acetabular cup implanted by a single surgeon. — The participant will undergo surgery using the hip prostheses and direct anterior surgical approach used by their surgeon-investigator. A patient-specific femoral guide, generated by the OPS™ Plan preoperatively, will be used during the surgical step of the femoral neck resection. These are not study specific procedures as the OPS™ Plan is already in use by the surgeon-investigator in their standard of care practice.

SUMMARY:
A prospective, non-randomized, single-center clinical study to determine the accuracy of a patient-specific instrument (OPS™) for delivering a planned femoral component anteversion and neck resection using a Direct Anterior Approach (DAA) in Total Hip Arthroplasy.

DETAILED DESCRIPTION:
Total Hip Replacement (THR) is the gold standard for treatment of severe arthritis of the hip as it relieves pain, restores function of the joint, and improves quality of life for patients. The restoration of hip mechanics can be influenced by the selected femoral stem design and also by choices made by the surgeon during the surgical implantation. The combination of femoral neck resection level and angle are key factors, particularly in cementless hip arthroplasty, in determining post-operative leg length and femoral anteversion. Historically, an estimation of prosthesis sizing and positioning has been made via a process of manual or digital templating either pre or intraoperatively using images of the implants positioned over the standard AP and lateral view hip x-rays taken in advance of surgery with generic instruments used during the surgery to execute the femoral head resection at the planned level. This process has a number of limitations. The OPS™ system utilizes detailed pre-operative imaging including a CT scan to generate a plan for the femoral neck resection level and angulation based on the anatomy of the individual patient. Following validation of this plan by the operating clinician, a patient specific femoral guide instrument is generated to help facilitate the reliable delivery of the planned resection intraoperatively. The purpose of this study will be to evaluate the use of the patient-specific femoral instrument in the hands of one surgeon using a protocol-specific choice of prosthesis combinations and one surgical approach. A total number of 100 subjects will be enrolled. Participants in this study will return for a single post-operative visit at 6 weeks to have x-rays taken and to enable any postoperative study hip-related complications recorded. Once this has been completed, participants will be routinely followed-up by their Orthopedic surgeon as required in accordance with the standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients who understand the conditions of the study and are willing to return to the clinical site at 2 weeks postoperatively.
* Patients of either gender who are between 21-85 years (inclusive) at the time of consent.
* Patients with a diagnosis of osteoarthritis (including post-traumatic osteoarthritis), rheumatoid arthritis or avascular necrosis and are considered by the Investigator to be clinically and medically suitable to undergo a primary total hip replacement.
* Patients who meet the indications and none of the contraindications listed in the Instructions for Use (IFU) supplied by the manufacturer for the femoral stem and acetabular cup to be implanted.
* Patients who meet the indications and none of the contraindications listed in the Instructions for Use (IFU) supplied by the manufacturer for OPS™ Femoral Plan and OPS™ Femoral Patient Specific Instruments.

Exclusion Criteria:

* Patients who are unable to provide informed consent.
* Patients who are unable to comply with all the required study procedures.
* Patients who are currently involved in any personal injury litigation, medical-legal or worker's compensations claims.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited from the surgeon's clinic. Those who meed the inclusion/exclusion criteria will be invited to enroll into the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-13 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the final osteotomy level compared to the selected OPS™ Plan | 2 weeks post-op (1 - 4 weeks post-op window)
  Accuracy of the final osteotomy level compared to the selected OPS™ Plan (+ or - 3 mm). Two standard of care postoperative x-rays taken at 2 weeks will be used to evaluate the positioning of the total hip prosthesis from the resultant level of resection of the femoral neck. This parameter will be measured in mm.

SECONDARY OUTCOMES:
Comparison of the femoral stem size implanted compared to the selected OPS™ Plan | Immediate postoperative
  Comparison of the femoral stem size implanted compared to the selected OPS™ Plan preoperatively (± 1 size). The femoral stem size used during the operation will be compared to the one selected by the OPS™ Plan. This parameter will be measured in units.
Comparison of the acetabular cup size implanted compared to the OPS™Plan | Immediate postoperative
  Comparison of the acetabular cup size implanted compared to the OPS™Plan preoperatively. The acetabular cup size used during the operation will be compared to the one selected by the OPS™ Plan. This parameter will be measured in mm.
Comparison of the femoral head size implanted compared to the selected OPS™ Plan | Immediate postoperative
  Comparison of the femoral head size implanted compared to the selected OPS™ Plan. This parameter will be measured in mm.
Measurement of any change in leg length / femoral head height compared to the preoperative OPS™ Plan | 2 weeks post-op (1 - 4 weeks post-op window)
  Measurement of any change in leg length / femoral head height compared to the preoperative OPS™ Plan (+ or - 5 mm). The postoperative leg length / femoral head height will be measured in mm and compared to the preoperative value.
Comparison of the acetabular cup orientation to the selected OPS™ Plan | 2 weeks post-op (1 - 4 weeks post-op window)
  Comparison of the acetabular cup orientation to the selected OPS™ Plan. The planned vs achieved acetabular cup orientation will be measured using 2D/3D registration software, in degrees.

CONTACTS AND LOCATIONS:
Overall Officials: Donald W Hohman, MD, Principal Investigator — Surgical Education & Research LLC
Locations (2):
- United States (2):
  - Texas Orthopaedic Associates, Dallas, Texas
  - Texas Orthopaedic Associates, Plano, Texas